CLINICAL TRIAL: NCT03327207
Title: Exploring Interactions Between Growth Hormone and the Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: 0132-17 RMB CTIL
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Children who receive Growth hormone treatment. Non Interventional
  Interventions: Other: Non Interventional
- Control group: Healthy children . Non Interventional
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional — Non Interventional

SUMMARY:
The goal of this study is to characterize the microbiome and metabolomics of children with Growth Hormone (GH) deficiency, prior GH treatment initiation and compare it to healthy children

ELIGIBILITY:
Inclusion Criteria:

* Children with GH deficiency

Exclusion Criteria:

* Turner syndrome
* End state renal disease (ESRD)
* Prader-Willi syndrome
* Systemic illness
* Antibiotics/Antifungal in the last 3m

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with GH deficiency
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Changes in the microbiome population following Growth hormone treatment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric endocrinology unit rambam medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided